CLINICAL TRIAL: NCT00404638
Title: Treatment of Enuresis Nocturna by Circular Muscle Exercise (Paula Method)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004192
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Monosymptomatic Enuresis Nocturna
Keywords: Enuresis Nocturna; Paula Method; Circular muscle exercise; Sphincter
MeSH Terms: conditions — Nocturnal Enuresis

INTERVENTIONS:
Drug: Desmopresin
Behavioral: Paula Method of Circular Muscle Exercise

SUMMARY:
Several treatment modalities for children suffering from monosymptomathic nocturnal enuresis are available including drugs, alarms, acupuncture, pelvic floor training and biofeedback. The aim of this study is to to test if Paula Method (circular muscle exercise) can be an another treatment modality.

DETAILED DESCRIPTION:
Paula method is based on circular muscle exercises. The theory behind the Paula method is that all sphincters in the human body work simultaneosly, mutually affecting one another possibly mediated by "oscillation" of the spinal cord. According to this theory, exercising the ring muscles in a certain area of the body will result in strengthening the circular muscles in other areas. This method was found to to be efficacious for treatment of urinary stress incontinence in women.

ELIGIBILITY:
Inclusion Criteria:

1. age- 7 to 15 years old suffering from monosymptomatic enuresis nocturna
2. informed consent

Exclusion Criteria:

1. UTI
2. neurological diseases or syndromes
3. metabolic disesaes
4. congenital disease or malformation of the urinary tract

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40
Dates: Start 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Herman A Cohen, MD, Principal Investigator — Schneider Children Hospital , Israel
Locations (2):
- Israel (2):
  - Campus Golda Hospital, Petah Tikva
  - Campus Rabin, Petah Tikva

REFERENCES:
- [Derived] Caldwell PH, Codarini M, Stewart F, Hahn D, Sureshkumar P. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2020 May 4;5(5):CD002911. doi: 10.1002/14651858.CD002911.pub3. PMID 32364251